CLINICAL TRIAL: NCT02888223
Title: Pharmacokinetic Comparison of SCT800 (B-domain Deleted Recombinant Factor VIII) With Xyntha in Previously Treated Patients With Hemophilia A: a Phase I, Open-label, Randomized, Crossover Study
Brief Title: Pharmacokinetic Study of SCT800 in Previously Treated Patients With Hemophilia A
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCT800HA1
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): a single dose administration of SCT800 followed by Xyntha (50 IU.kg-1, based upon the manufacturer's labeled potency)
  Interventions: Biological: SCT800; Biological: Xyntha
- Group B (Experimental): a single dose administration of Xyntha followed by SCT800(50 IU.kg-1, based upon the manufacturer's labeled potency)
  Interventions: Biological: SCT800; Biological: Xyntha

INTERVENTIONS:
Biological: SCT800
  Other Names: Recombinant human coagulation factor VIII
Biological: Xyntha
  Other Names: Antihemophilic Factor (Recombinant), Plasma/Albumin-Free

SUMMARY:
Participants will be assigned to A or B groups with a scale of 1:1 based on a prospectively randomized treatment-sequence assignment, i.e. infuse SCT800 followed by Xyntha (group A), or the alternate sequence (group B). All participants who completed the SCT800HA1 study will enter the efficacy and safety study (Protocol No.: SCT800HA3).

ELIGIBILITY:
Inclusion Criteria:

* 12 to 65 years old;
* The activity of the coagulation factor VIII (FVIII:C) ≤2%, and was previously treated with FVIII concentrate(s) for a minimum of 50 exposure days (EDs) prior to study entry
* Non-bleeding state (No clinical manifestations of active hemorrhage);
* Negative assays for FVIII inhibitors (<0.6 BU/mL);
* The platelet count is normal；
* Normal prothrombin time or INR ≤1.5；
* Given informed consent

Exclusion Criteria:

* Hypersensitivity to recombinant coagulation factor VIII concentrate or any of the excipients ;allergic to heterologous proteins (e.g. murine, bovine or hamster origin);
* Family history or history of FVIII inhibitors (≥0.6 Bethesda Units [BU] mL-1);
* Received an infusion of any FVIII for on-demand therapy or prophylaxis within 4 days prior to study entry (including rFVIII, plasma-derived factor VIII [pdFVIII], cryoprecipitate and whole blood);
* Significant hepatic or renal impairment (ALT and AST ≥2×ULN; BUN and Cr≥2×ULN);
* HIV seropositive;
* Abnormal hemostasis from causes other than hemophilia A；
* Patients with severe heart disease, including myocardial infarction, heart failure (III or higher level);
* Patients who received any anticoagulant or antiplatelet therapy within one week (including NSAIDs) or need to receive an anticoagulant or antiplatelet therapy during the period of clinical trials;
* Alcoholism, drug abuse, mental disorders and mental retardation;
* Elective surgery planned during the process of study;
* Patients who previously participated in the other clinical trials prior to study entry;
* The patient or parent/legal guardian is unable or unwilling to sign an informed consent form or to comply with the requirements of clinical protocol;
* Other conditions confirmed by the researchers, resulting in that patients are unable to benefit from clinical observation;

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-02 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Incremental Recovery (K-value) | 1hour after the end of the infusion
  One-stage aPTT Assay
Area Under the Plasma Concentration Versus Time Curve From 0 to 48 Hours (AUClast) | 48 hours after the end of the infusion
  One-stage aPTT Assay
Elimination Phase Half-life (t1/2) | 48 hours after the end of the infusion
  One-stage aPTT Assay
Factor VIII (FVIII) Clearance (CL) | 48 hours after the end of the infusion
  One-stage aPTT Assay

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Versus Time Curve From 0 to Infinity (AUC∞) | 48 hours after the end of the infusion
  One-stage aPTT Assay
FVIII Maximum Plasma Concentration (Cmax) | 3 hours after the end of the infusion
  One-stage aPTT Assay
Mean Residence Time (MRT) | 48 hours after the end of the infusion
  One-stage aPTT Assay
Volume of Distribution at Steady State (Vss) | 48 hours after the end of the infusion
  One-stage aPTT Assay
Incidence of inhibitors | 72 hours after the end of the infusion
AEs related to SCT800 during treatment and observation of the clinical study | 48 hours after the end of the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Xie lan Zhao, PhD, Principal Investigator — Xiangya Hospital of Centre-South University, Changsha, China
Locations (1):
- Xiangya Hospital of Centre-South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No